CLINICAL TRIAL: NCT06899932
Title: Survival Study of the Genutech® Total Knee Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Hospital de Sant Rafael (Other)
Responsible Party: Sponsor
Other Study IDs: PR-2021-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective cohort sudy of patients undergoing a Genutech® total knee arthroplasty

DETAILED DESCRIPTION:
A prospective cohort study will be performed collecting patient's data before and after the total knee arthroplasty surgical procedure at one, five and ten years. The main goal of this work is to prospectively study the results obtained with the implantation of the knee prosthesis currently used in the Orthopaedic Service of Sant Rafael Hospital of Barcelona (Genutech®). The main outcome of the study is the survival of the implant, that is, having no revision surgeries in the follow-up. The secondary objective is the clinical and radiological evaluation of the implants measured by outcome measueres: Oxford Knee Score (OKS), SF12 questionnaire and WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionaire. OKS and SF12 scores are higher with good results and lower with bad results. WOMAC expresses results the other way around.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with knee osteoarthritis that had not responded to conservative treatment
* capable of providing informed consent
* patients who receive a Genutech® total knee prosthesis at the investigators' Institution.

Exclusion Criteria:

* having received a prior total knee arthroplasty in the same joint
* inability to provide informed consent
* not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the investigators' Institution by Primary Care centres to receive Orthopaedic care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients without revision surgery | 5 and 10 years
  the main goal is to determine the implant survival, that is, having no revision during follow-up. The number of patients requiring revision will be compared to the total of patients included in the study.

SECONDARY OUTCOMES:
Oxford Knee Score | one, 5 and 10 years
  Clinical evaluation with Patient Reported Outome Measures (PROMs): Oxford Knee Score (OKS). OKS score is higher with good results and lower with bad results.
SF12 questionnaire | 1, 5 and 10 years postoperatively
  Clinical evaluation with Patient Reported Outome Measures (PROMs): SF12 questionnaire. SF12 scores are higher with good results and lower with bad results.
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionaire | One, 5 and 10 years
  Clinical evaluation with Patient Reported Outome Measures (PROMs): WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) questionaire. WOMAC scores are higher with bad results and lower with good results.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Rafael, Barcelona, Barcelona, Spain